CLINICAL TRIAL: NCT01826214
Title: A Phase II Multi-center, Open Label, Randomized Study to Assess Safety and Efficacy of Two Different Schedules of Oral LDE225 in Adult Patients With Relapsed/Refractory or Untreated Elderly Patients With Acute Leukemia
Brief Title: Study of Efficacy and Safety of LDE225 in Adult Patients With Relapsed/Refractory Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X2203
Record Dates: First submitted 2013-03-25; First posted 2013-04-08 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Acute Leukemias
Keywords: acute myeloid leukemia; AML; acute lymphoblastic leukemia; ALL; leukemia; acute; LDE225; adult patients; relapsed/refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Recurrence | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDE225-400 (Experimental): Patients who were randomized to Schedule A, and received 400 mg LDE225 twice daily for the first two weeks only and then after two weeks, received 800 mg LDE225 once daily until disease progression, toxicity, withdrawal of consent, death, discretion of the investigator or early termination of the study.
  Interventions: Drug: LDE225
- LDE225-800 (Experimental): Patients who were randomized to Schedule B, received 800 mg LDE225 once daily until disease progression, toxicity, withdrawal of consent, death, discretion of the investigator or early termination of the study.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225 will be supplied as 200 mg capsules by Novartis. Patients will receive study treatment on an outpatient basis. LDE225 will be dispensed every two weeks for the first four weeks and at the start of every four weeks thereafter, as needed.

SUMMARY:
The study will evaluate the efficacy, safety and tolerability of two dosing schedules of LDE225 in patients with relapsed/refractory acute leukemia or elderly patients with untreated acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have relapsed or primary refractory non-M3 acute myeloid leukemia or relapsed or refractory non-T-cell acute lymphoblastic leukemia or untreated acute myeloid leukemia in elderly patients.
* Performance status of 0, 1 or 2 per WHO classification.
* Adequate renal and liver function.
* Adequate blood creatine kinase value (CK < 1.5ULN)

Exclusion Criteria:

* Allogeneic stem cell transplantation within the last 4 months and/or active graft versus host disease requiring systemic immunosuppressant therapy, or autologous stem cell transplantation within the last 4 weeks.
* Patient for which immediate allogeneic stem cell transplantation is the treatment of choice.
* Pregnant or nursing (lactating) women.
* Active CNS leukemic involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Duke University Medical Center SC-5, Durham, North Carolina, United States
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Prahran, Victoria
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Yvoir
- Novartis Investigative Site, Montreal, Quebec, Canada
- Germany (4):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Debrecen, Hungary
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Trondheim
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 patients were randomized but only 34 patients received at least one dose of study drug in the LDE225-800 (schedule B ) arm.
Groups:
- LDE225-400: Patients who were randomized to Schedule A, and received 400 mg LDE225 twice daily for the first two weeks only and after two weeks, received 800 mg LDE225 once daily until disease progression, toxicity, withdrawal of consent, death, discretion of the investigator or early termination of the study.
Period: Overall Study
Arm/Group | LDE225-400 | LDE225-800
Started | 35 | 34 (35 patients were randomized but only 34 patients received at least one dose of study drug)
Untreated | 0 (Untreated = did not receive study drug) | 1 (Untreated = did not receive study drug)
Treated | 35 (Treated = received at least one dose of study drug) | 34 (Treated = received at least one dose of study drug)
Completed | 0 | 0
Not Completed | 35 | 34
Not completed — Adverse Event | 7 | 6
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Progressive disease | 22 | 21
Not completed — Study terminated by Sponsor | 0 | 1
Not completed — Subject/guardian decision | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): comprised of all patients who were randomized to a study treatment.
  According to the intent-to-treat principle, patient data were analyzed according to the treatment to which they had been randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225-400 | LDE225-800 | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (12.31) | 67.7 (11.65) | 66.5 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission (CR)
Description: Complete Response (CR) was based on the International Working Group (IWG) criteria based on weekly peripheral blood count measurements and bone marrow biopsy/aspiration collection. Efficacy assessments were performed to determine CR. A treatment cycle was defined as 4 weeks. The outcome measure for the study is based on standardized response criteria as defined by the International Working Group (IWG) for AML. The IWG was established by a group of investigators interested in the design and conduct of clinical trials in acute myeloid leukemia (AML). The criteria established by this group (a set of recommendations for response assessment) are well established, endorsed by major institutions and Health Authorities, and are widely used in clinical trials. No statistical analysis was planned for this primary outcome.
Time Frame: at screening, every week up to Week 9, every 2 weeks thereafter until CR, every 4 weeks after CR up to 24 months
Population: Full analysis set (FAS): comprised of all patients who were randomized to a study treatment.
  According to the intent-to-treat principle, patient data were analyzed according to the treatment to which they had been randomized. No statistical analysis were reported in this study.
Measure: Number; unit: Participants
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

2. Primary Outcome: Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: The other primary efficacy endpoint was CRi based on the International Working Group (IWG) criteria based on weekly peripheral blood count measurements and bone marrow biopsy/aspiration collection. Efficacy assessments were performed to determine CRi. A treatment cycle was defined as 4 weeks. No statistical analysis was planned for this primary outcome.
Time Frame: within 3 days after clearance of blasts from peripheral blood (PB), monthly thereafter until CR or reappearance of blasts in the PB, after CR every other month until discontination up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 35 | 35
Participants | 1 | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was the rate of complete remission (CR), complete remission with incomplete blood count recovery (CRi) or partial response (PR) according to IWG criteria. CR, CRi or PR will be assessed through bone marrow biopsy/aspirate and peripheral blood blasts counts.
Time Frame: Every 8 weeks for the first 6 months and every 12 weeks until 53 weeks after the last patient is enrolled or until relapse up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 35 | 35
Participants | 1 | 0

4. Secondary Outcome: Parmacokintics (PK) Parameter: Cmax
Description: Cmax is the maximum observed plasma concentration after drug administration.The PK parameters were determined in plasma using non-compartmental methods. A PK sample was excluded from analyses if the patient vomited within the first 4 hours following the last oral dose of study drug. Other PK samples were excluded as deemed appropriate by the pharmacokineticist. Cmax was derived from the PK concentrations collected at 0, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose on W1D1 and W9D1. The PK concentration at each time point is not an endpoint in the protocol, but these concentrations are used to derive the PK parameters.
Time Frame: Week 1 Day 1, Week 9 Day 1
Population: Pharmacokinetic analysis set (PAS): consisted of all patients who received at least one dose of sonidegib and provided at least one evaluable PK blood sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 29 | 33
ng/mL
  Week 1 Day 1 | 237 (158) | 343 (275)
  Week 9 Day 1(n: 7, 7) | 1640 (612) | 1500 (874)

5. Secondary Outcome: Parmacokintics (PK) Parameter: Tmax
Description: Tmax is the time to reach Cmax. The PK parameters were determined in plasma using non-compartmental methods. A PK sample was excluded from analyses if the patient vomited within the first 4 hours following the last oral dose of study drug. Other PK samples were excluded as deemed appropriate by the Pharmacokineticist. Tmax was derived from the PK concentrations collected at 0, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose on W1D1 and W9D1. The PK concentration at each time point is not an endpoint in the protocol, but these concentrations are used to derive the PK parameters.
Time Frame: Week 1 Day 1,Week 9 Day 1
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 29 | 33
hr
  Week 1 Day 1 | 2.13 (NA) [1.00 to 8.08] | 2.12 (NA) [1.00 to 8.00]
  Week 9 Day 1 (n: 7, 7) | 1.88 (NA) [1.12 to 8.13] | 2.02 (NA) [0.00 to 23.3]

6. Secondary Outcome: Parmacokintics (PK) Parameter: AUC0-8h
Description: AUC0-8h is the area under the concentration-time curve from time zero to 8 hours. The PK parameters were determined in plasma using non-compartmental methods. A PK sample was excluded from analyses if the patient vomited within the first 4 hours following the last oral dose of study drug. Other PK samples were excluded as deemed appropriate by the Pharmacokineticist. AUC0-8h was derived from the PK concentrations collected at 0, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose on W1D1 and W9D1. The PK concentration at each time point is not an endpoint in the protocol, but these concentrations are used to derive the PK parameters.
Time Frame: Week 1 Day 1,Week 9 Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 27 | 33
ng*hr/mL
  Week 1 Day1 | 988 (542) | 1560 (1230)
  Week 9 Day1 (n: 7, 7) | 9750 (2830) | 7910 (5090)

7. Secondary Outcome: Parmacokintics (PK) Parameter: AUC0-24h
Description: AUC0-24 is the area under the concentration-time curve from time zero to 24 hours done only on 800 mg once a day schedule. The PK parameters were determined in plasma using non-compartmental methods. A PK sample was excluded from analyses if the patient vomited within the first 4 hours following the last oral dose of study drug. Other PK samples were excluded as deemed appropriate by the Pharmacokineticist. AUC0-24h was derived from the PK concentrations collected at 0, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose on W1D1 and W9D1. The PK concentration at each time point is not an endpoint in the protocol, but these concentrations are used to derive the PK parameters.
Time Frame: Week 1 Day 1,Week 9 Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LDE225-400 | LDE225-800
Number analyzed (Participants) | 7 | 32
ng*hr/mL
  Week 1 Day 1 | 0 (0) | 3110 (2620)
  Week 9 Day 1 (n: 7, 6) | 26500 (6650) | 24000 (11500)

ADVERSE EVENTS:
Arm/Group | LDE225-400 | LDE225-800
Serious Adverse Events (participants affected / at risk) | 25/35 | 25/34
Other Adverse Events (participants affected / at risk) | 35/35 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225-400 (N=35) | LDE225-800 (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GINGIVAL HYPERTROPHY (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 2 | 1
FATIGUE (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 4
ANAL ABSCESS (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 2 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 3
SEPSIS (Infections and infestations) | 2 | 4
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 | 2
MYOGLOBIN BLOOD INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEUKAEMIC INFILTRATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1
QUADRIPLEGIA (Nervous system disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
IDIOPATHIC PNEUMONIA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225-400 (N=35) | LDE225-800 (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 6
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 6 | 8
DIARRHOEA (Gastrointestinal disorders) | 7 | 8
DYSPEPSIA (Gastrointestinal disorders) | 3 | 3
DYSPHAGIA (Gastrointestinal disorders) | 0 | 2
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 3
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 3
MOUTH ULCERATION (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 11 | 10
ORAL DISORDER (Gastrointestinal disorders) | 2 | 0
ORAL PAIN (Gastrointestinal disorders) | 1 | 3
VOMITING (Gastrointestinal disorders) | 7 | 12
ASTHENIA (General disorders) | 1 | 2
CHILLS (General disorders) | 2 | 0
FATIGUE (General disorders) | 8 | 10
FEELING COLD (General disorders) | 2 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 3
MALAISE (General disorders) | 1 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 4 | 5
PAIN (General disorders) | 0 | 3
PYREXIA (General disorders) | 7 | 10
INFECTION (Infections and infestations) | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 1 | 2
ORAL HERPES (Infections and infestations) | 2 | 1
SKIN INFECTION (Infections and infestations) | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 3
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2
FALL (Injury, poisoning and procedural complications) | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 8 | 7
BLOOD CREATININE INCREASED (Investigations) | 1 | 5
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 2
MYOGLOBIN BLOOD INCREASED (Investigations) | 2 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 2
PLATELET COUNT DECREASED (Investigations) | 2 | 2
WEIGHT DECREASED (Investigations) | 2 | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 | 5
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 6
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 8 | 5
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 8
MYOPATHY (Musculoskeletal and connective tissue disorders) | 2 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 4
DIZZINESS (Nervous system disorders) | 2 | 5
DYSGEUSIA (Nervous system disorders) | 3 | 5
HEADACHE (Nervous system disorders) | 3 | 5
ANXIETY (Psychiatric disorders) | 4 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 4 | 0
INSOMNIA (Psychiatric disorders) | 2 | 2
DYSURIA (Renal and urinary disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 6
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 6
RASH (Skin and subcutaneous tissue disorders) | 4 | 2
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 | 0
HAEMATOMA (Vascular disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 0 | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Only 34 of the 35 patients in the LDE225 800 mg once daily arm received at least dose of study drug were analyzed for safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.